CLINICAL TRIAL: NCT07004049
Title: TREAT-GNB [CR-GNB]
Brief Title: Optimising TREATment for Severe Gram-Negative Bacterial Infections
Acronym: TREAT-GNB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: The University of Queensland (Other); European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Responsible Party: Principal Investigator, Mo Yin, Consultant / Adjunct Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ADVANCE-ID 24003
Record Dates: First submitted 2025-04-29; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Bloodstream Infection; Ventilator Associated Bacterial Pneumonia; Hospital Acquired Bacterial Pneumonia; Carbapenem Resistant Bacterial Infection; Multidrug Resistance
MeSH Terms: conditions — Sepsis | interventions — Colistin; Polymyxin B; Sulbactam; Meropenem; avibactam, ceftazidime drug combination; Fosfomycin; Aztreonam; meropenem and vaborbactam; Cefiderocol; ceftolozane, tazobactam drug combination

STUDY DESIGN:
Intervention Model Description: The backbone domain is a multi-arm antibiotic treatment intervention with a personalisable randomisation list. It adopts the "Personalised Randomised Controlled Trial" (PRACTical) design, which allows each participant to be randomised between a personalised randomisation list of treatments that are suitable for them. Each patient randomisation list ("personalised randomisation list") may be tailored based on their kidney function, pathogen genotype, pathogen antibiotic susceptibility and physician preference. Potential participants may be enrolled and randomised if they are eligible for at least two antibiotic options in the site randomisation list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Colistin/Polymyxin B + Sulbactam (Active Comparator)
  Interventions: Drug: Colistin/Polymyxin B + Sulbactam
- Colistin/Polymyxin B + Tigecycline/Eravacycline (Active Comparator)
  Interventions: Drug: Colistin/Polymyxin B + Tigecycline/Eravacycline
- Colistin/Polymyxin B + Meropenem (Active Comparator)
  Interventions: Drug: Colistin/Polymyxin B + Meropenem
- Ceftazidime-avibactam + Sulbactam (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam + Sulbactam
- Ceftazidime-avibactam + Fosfomycin (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam + Fosfomycin
- Ceftazidime-avibactam (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam
- Ceftazidime-avibactam + Aztreonam (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam + Aztreonam
- Ceftazidime-avibactam + Colistin/Polymyxin B (Active Comparator)
  Interventions: Drug: Ceftazidime-avibactam + Colistin/Polymyxin B
- High-dose meropenem (Active Comparator)
  Interventions: Drug: High-dose meropenem
- Meropenem + Fosfomycin (Active Comparator)
  Interventions: Drug: Meropenem + Fosfomycin
- Meropenem-vaborbactam (Active Comparator)
  Interventions: Drug: Meropenem-vaborbactam
- Cefiderocol (Active Comparator)
  Interventions: Drug: Cefiderocol
- Ceftolozane-tazobactam (Active Comparator)
  Interventions: Drug: Ceftolozane-tazobactam
- Ceftolozane-tazobactam + Meropenem (Active Comparator)
  Interventions: Drug: Ceftolozane-tazobactam + Meropenem

INTERVENTIONS:
Drug: Colistin/Polymyxin B + Sulbactam — For carbapenem-resistant Acinetobacter infections in China, Malaysia, Thailand and Singapore
  Arms: Colistin/Polymyxin B + Sulbactam
Drug: Colistin/Polymyxin B + Tigecycline/Eravacycline — For carbapenem-resistant Acintobacter, carbapenem-resistant Enterobacterales infections in China, Malaysia, Thailand and Singapore
  Arms: Colistin/Polymyxin B + Tigecycline/Eravacycline
Drug: Colistin/Polymyxin B + Meropenem — For carbapenem-resistant Pseudomonas aeruginosa, carbapenem-resistant Enterobacterales infections in China, Malaysia and Singapore
  Arms: Colistin/Polymyxin B + Meropenem
Drug: Ceftazidime-avibactam + Sulbactam — For carbapenem-resistant Acinetobacter infections in China, Malaysia, Thailand, Singapore and Australia.
  Arms: Ceftazidime-avibactam + Sulbactam
Drug: Ceftazidime-avibactam + Fosfomycin — For carbapenem-resistant Pseudomonas aeruginosa, carbapenem-resistant Enterobacterales infections in Malaysia, Thailand and Singapore
  Arms: Ceftazidime-avibactam + Fosfomycin
Drug: Ceftazidime-avibactam — For carbapenem-resistant Pseudomonas aeruginosa, carbapenem-resistant Enterobacterales infections in China, Malaysia, Thailand, Singapore, Europe and Australia.
  Arms: Ceftazidime-avibactam
Drug: Ceftazidime-avibactam + Aztreonam — For carbapenem-resistant Enterobacterales infections in China, Malaysia, Thailand, Singapore, Europe and Australia.
  Arms: Ceftazidime-avibactam + Aztreonam
Drug: Ceftazidime-avibactam + Colistin/Polymyxin B — For carbapenem-resistant Pseudomonas aeruginosa in China, Malaysia, Thailand, Singapore and Europe.
  Arms: Ceftazidime-avibactam + Colistin/Polymyxin B
Drug: High-dose meropenem — For carbapenem-resistant Enterobacterales infection in Europe
  Arms: High-dose meropenem
Drug: Meropenem + Fosfomycin — For carbapenem-resistant Enterobacterales in Europe
  Arms: Meropenem + Fosfomycin
Drug: Meropenem-vaborbactam — For carbapenem-resistant Enterobacterales infection in Europe
  Arms: Meropenem-vaborbactam
Drug: Cefiderocol — For carbapenem-resistant Pseudomonas aeruginosa, carbapenem-resistant Enterobacterales infections in Europe and Australia.
  Arms: Cefiderocol
Drug: Ceftolozane-tazobactam — For carbapenem-resistant Pseudomonas aeruginosa in Europe and Australia.
  Arms: Ceftolozane-tazobactam
Drug: Ceftolozane-tazobactam + Meropenem — For carbapenem-resistant Pseudomonas aeruginosa in Europe.
  Arms: Ceftolozane-tazobactam + Meropenem

SUMMARY:
TREAT-GNB is an innovative trial to expedite the evaluation of various antibiotic choices and treatment strategies for severe multidrug-resistant Gram-negative bacterial infections, specifically bloodstream and lower respiratory tract infections. This approach combines platform trial elements with adaptive clinical designs to streamline the evaluation of various treatment options and optimise resource utilisation. The overall aim of the TREAT-GNB platform trial is to identify interventions that improve survival in patients with severe infections due to Gram-negative bacteria.

In the CR-GNB silo of TREAT-GNB, the primary objective is to quantify the effect on all-cause mortality at 28 days of a range of interventions in patients with bloodstream infections, ventilator-associated pneumonia, and hospital-acquired pneumonia caused by CR-GNB.

ELIGIBILITY:
Inclusion Criteria:

A: Bloodstream infections

a) Suitable for at least 2 antibiotic regimens in the site randomisation list

1. Growth of Gram-negative bacilli identified from blood culture(s)
2. Receiving or planning to receive intravenous antibiotics
3. Expected time from blood culture sampling to randomisation is ≤ 96 hours.

OR

B: Ventilator-associated pneumonia / hospital-acquired pneumonia a) Suitable for at least 2 antibiotic regimens in the site randomisation list b) Infection syndrome definitions^( (US Centers for Disease Control and Prevention National Healthcare Safety Network)3: i) At least one of the following:

1. temperature > 38 °C
2. white blood cell count ≥ 12,000 cells/mm3 (12 x 109/L, 12 x 103/µL) or ≤ 4,000 cells/mm3 (4 x 109/L, 4 x 103/µL)
3. altered mental status with no other causes in > 70 years old; AND ii) Two or more chest imaging tests demonstrating at least one of the following:

1) new and progressive OR progressive and persistent infiltrate 2) new and persistent OR progressive and persistent consolidation 3) new and persistent OR progressive and persistent cavitation; AND iii) At least two of the following:

1. new onset of purulent sputum, or change in character of sputum, or increased respiratory secretions, or increased in suctioning requirements
2. new onset or worsening tachypnoea or dyspnoea
3. rales or bronchial breath sounds
4. worsening gas exchange defined by oxygen desaturations (e.g., PaO2/FiO2 < 240), increased oxygen requirements or increased ventilation demand.

   c) Hospital admission > 48 hours d) Predominant growth of Gram-negative bacilli identified from respiratory tract specimen(s)*; e) Receiving or planning to receive intravenous antibiotics f) Expected time from respiratory culture sampling to randomisation is ≤ 96 hours

   AND

   C: CR-GNB antibiotic backbone domain

   a) Gram-negative bacilli belonging to Acinetobacter baumannii-calcoaceticus complex, Pseudomonas aeruginosa or Enterobacterales b) Carbapenem resistance in isolate detected - i) Phenotypically via conventional microbiology testing: meropenem / imipenem / ertapenem resistance; OR ii) Genotypically via PCR or next generation sequencing: presence of genes associated with carbapenemase production (eg. blaNDM, blaKPC, blaIMP, blaIMI, blaVIM, blaOXA-48-like).

   Exclusion Criteria:
   1. Treating team deems enrolment in the study is not in the best interest of the patient
   2. Patient is on end-of-life care
   3. Patient is incarcerated in a correctional facility
   4. Participation in any interventional study activities outlined in the TREAT-GNB study within the last 90 days
   5. Pregnant women and children

      OR
   6. Polymicrobial bloodstream infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 28 days post-randomisation
  28-day all-cause mortality after randomisation

SECONDARY OUTCOMES:
Clinical outcome | 14, 60 and 90 days post-randomisation
  All-cause mortality at 14, 60 and 90 days after randomisation
Clinical outcome | 90 days post-randomisation
  Proportion of patients with infection relapse or reinfection within 90 days after randomisation
Clinical outcome | 28 days post-randomisation
  Length of mechanical ventilation in the intensive care within 28 days after randomisation
Clinical outcome | 90 days post-randomisation
  All cause re-admission into an acute care hospital within 90 days after randomisation
Clinical outcome | 28 days post-randomisation
  Proportion of patients that develop Kidney Disease Improving Global Outcomes (KDIGO) acute kidney injury within 28 days after randomisation
Clinical outcome | 28 days post-randomisation
  Proportion of patients that develop Clostridioides difficile or antibiotic-related diarrhea within 28 days after randomisation
Clinical outcome | 28 and 90 days post-randomisation
  Proportion of participants who have returned to their usual level of function at day 28 and 90 as determined by whether the modified functional bloodstream infection score (FBIS) remained the same or improved from baseline
Clinical outcome | 28 days post-randomisation
  Composite outcome measure defined by Desirability of Outcome Ranking (DOOR) at 28 days after randomisation
Clinical outcome | 14 days post-randomisation
  Sequential Organ Failure Assessment (SOFA) Score (0 to 24) improvement between baseline and 14 days after randomisation
Clinical outcome | 14 days post-randomisation
  Clinical response at 14 days after randomisation (Binary outcome: Improved or not improved, determined using 1. Temperature < 38°C for 48hours, and 2. Systolic blood pressure >90mmHg without inotropes)
Clinical outcome | 14, 28 and 90 days post-randomisation
  Clinical cure at 14, 28 and 90 days after randomisation (binary outcome: cure or no cure, as defined in the INHALE trial for VAP/HAP and in Yahav et al. trial for BSI)
Health economics outcomes | 28 days post-randomisation
  Length of continuous stay in the intensive care from the hospital which the participant was recruited within 28 days after randomisation
Health economics outcomes | 28 days post-randomisation
  Length of continuous stay in the hospital which the participant was recruited within 28 days after randomisation
Health economics outcomes | 28 days post-randomisation
  Days of antibiotic use within 28 days after randomisation
Health economics outcomes | 28 and 90 days post-randomisation
  Functional outcome at 28 and 90 days after randomisation (measured using EQ-5D-3L: https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-3l/)

CONTACTS AND LOCATIONS:
Locations (41):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane
- China (3):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital, Xi'an Jiang Tong University, Xi'an
  - Xuzhou First People's Hospital, Xuzhou
- American University of Beirut Medical Center, Beirut, Lebanon
- Malaysia (5):
  - Queen Elizabeth I, Kota Kinabalu, Sabah
  - Queen Elizabeth II, Kota Kinabalu, Sabah
  - Miri Sarawak Hospital, Miri, Sarawak
  - Ampang Hospital, Ampang, Selangor
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
- Hamad Medical Corporation, Doha, Qatar
- King Saud bin Abdulaziz University for Health Sciences, Riyadh, Saudi Arabia
- National University Hospital, Singapore, Singapore, Singapore
- Helen Joseph Hospital, Johannesburg, South Africa
- Spain (21):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital del Mar Barcelona, Barcelona
  - Hospital Universitario Bellvitge, Barcelona
  - Hospital Universitario Reina Sofía Córdoba, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Álvaro Cunqueiro, Pontevedra
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Thailand (3):
  - Phramongkutkloa Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiangmai University, Chiang Mai
- İstanbul Medipol Üniversitesi, Istanbul, Turkey (Türkiye)
- Dubai Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data

REFERENCES:
- [Background] Niederman MS, Alder J, Bassetti M, Boateng F, Cao B, Corkery K, Dhand R, Kaye KS, Lawatscheck R, McLeroth P, Nicolau DP, Wang C, Wood GC, Wunderink RG, Chastre J. Inhaled amikacin adjunctive to intravenous standard-of-care antibiotics in mechanically ventilated patients with Gram-negative pneumonia (INHALE): a double-blind, randomised, placebo-controlled, phase 3, superiority trial. Lancet Infect Dis. 2020 Mar;20(3):330-340. doi: 10.1016/S1473-3099(19)30574-2. Epub 2019 Dec 19. PMID 31866328
- [Background] Yahav D, Franceschini E, Koppel F, Turjeman A, Babich T, Bitterman R, Neuberger A, Ghanem-Zoubi N, Santoro A, Eliakim-Raz N, Pertzov B, Steinmetz T, Stern A, Dickstein Y, Maroun E, Zayyad H, Bishara J, Alon D, Edel Y, Goldberg E, Venturelli C, Mussini C, Leibovici L, Paul M; Bacteremia Duration Study Group. Seven Versus 14 Days of Antibiotic Therapy for Uncomplicated Gram-negative Bacteremia: A Noninferiority Randomized Controlled Trial. Clin Infect Dis. 2019 Sep 13;69(7):1091-1098. doi: 10.1093/cid/ciy1054. PMID 30535100
- [Background] McNamara JF, Harris PNA, Chatfield MD, Lorenc P, Paterson DL. Measuring patient-centred long-term outcome following a bloodstream infection: a pilot study. Clin Microbiol Infect. 2020 Feb;26(2):257.e1-257.e4. doi: 10.1016/j.cmi.2019.10.011. Epub 2019 Oct 23. PMID 31654791
- [Background] Evans SR, Rubin D, Follmann D, Pennello G, Huskins WC, Powers JH, Schoenfeld D, Chuang-Stein C, Cosgrove SE, Fowler VG Jr, Lautenbach E, Chambers HF. Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR). Clin Infect Dis. 2015 Sep 1;61(5):800-6. doi: 10.1093/cid/civ495. Epub 2015 Jun 25. PMID 26113652
- [Background] Walker AS, White IR, Turner RM, Hsu LY, Yeo TW, White NJ, Sharland M, Thwaites GE. Personalised randomised controlled trial designs-a new paradigm to define optimal treatments for carbapenem-resistant infections. Lancet Infect Dis. 2021 Jun;21(6):e175-e181. doi: 10.1016/S1473-3099(20)30791-X. Epub 2021 Apr 21. PMID 33894130